CLINICAL TRIAL: NCT03038295
Title: Safety and Efficacy of Propranolol Treatment in Newborns With Retinopathy of Prematurity:a Prospective Cohort Study
Brief Title: a Prospective Cohort Study for Propranolol Treatment in Retinopathy of Prematurity
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangdong Women and Children Hospital (Other)
Responsible Party: Principal Investigator, Nie Chuan, Vice director of Department of Neonatology, Guangdong Women and Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lqiong
Record Dates: First submitted 2017-01-19; First posted 2017-01-31 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; propranolol; ROP
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Propranolol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- oral propranol group (Experimental): Enrolled preterm newborns will receive oral propranolol 0.25mg/kg daily(every 24 hours).
  The treatment will be started as soon as the diagnosis of stage 1 or 2 ROP without plus is made and will be continue until the development of retinal vascularization is completed, but no more than 90 days.
  Interventions: Drug: Propranolol
- oral placebo group (Placebo Comparator): Enrolled preterm newborns will receive oral normal saline 0.25mg/kg daily(every 24 hours) and other disposals will be done similarily to the oral propranol group.
  Interventions: Drug: placebo
- eye drop propranol group (Experimental): Enrolled preterm newborns will receive propranolol as ophthalmic solution (0.2%). 3 microdrops of 6 microliters (μL) propranolol solution (= 6 μg propranolol/microdrop) will be topically applied with a calibrated pipette,in each eye, four times daily (every 6 hours) .
  The treatment will be started as soon as the diagnosis of stage 1 or 2 ROP without plus is made and will be continue until the development of retinal vascularization is completed, but no more than 90 days.
  Interventions: Drug: Propranolol
- eye drop placebo group (Placebo Comparator): Enrolled preterm newborns will receive placebo as ophthalmic solution in the same way of eye drop propranolol and other disposals will be done similarily to the eye drop propranol group.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Propranolol — Oral propranolol:0.25mg/kg daily(every 24 hours)；Eye drop propranolol(0.2%):3 microdrops,in each eye, four times daily (every 6 hours) .Both administration routes will be discontinued until retinal vascularization will be completed, but no more than 90 days.The study will be discontinued immediately in the presence of serious adverse effects attributable to the pharmacological actions of propranolol (severe hypotension, bradycardia or bronchospasm).In case of surgery or induction of anesthesia during the administration of propranolol, the drug should be discontinued at least 24 hours before surgery.In cases of severe hypotension or bradycardia may be administered one or more of the following drugs:Atropine.Isoproterenol hydrochloride (isoprenaline).Terlipressin.Glucagon In case of severe bronchospasm may be used salbutamol aerosol or salbutamol + ipratropium bromide. Betamethasone could be used for aerosol or systemic (intravenous or intramuscular).
  Arms: eye drop propranol group; oral propranol group
Drug: placebo — Oral/eye drop placebo will be taken in enrolled newborns. Other treatment will follow the standard treatment schedule of Early Treatment For Retinopathy Of Prematurity Cooperative Group.
  Other Names: normal saline
  Arms: eye drop placebo group; oral placebo group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of oral/local propranolol in preterm newborns who diagnosed as early phase of retinopathy of prematurity (ROP).

DETAILED DESCRIPTION:
The incidence of Retinopathy of Prematurity (ROP) in preterm newborns less than 1500g is about 60% in the developed countries around the world, while there are much more preterm newborns more than 1500g and 32 weeks gestational age with Retinopathy of Prematurity (ROP) had to be treated in the developing countries. ROP has listed top of the five causes lead to blindness in children, which seriously threated children's vision and quality of life.

The ablation of the retina with photocoagulation by laser or cryotherapy reduces the incidence of blindness by suppressing the neovascular phase of ROP. However, those Surgeries require anesthesia and some of them may result in complications such as apnea, neonatal necrotizing enterocolitis, sepsis, and hemorrhage of digestive tract. As a result, it's important to study an alternative non-surgical treatment method.

The development of ROP depends largely from vascular endothelial growth factor (VEGF). The reduction of VEGF expression in the neovascular phase might prevent destructive neovascularization in ROP.

Propranolol is a kind of beta-adrenergic receptor (β-AR) which can inhibit the expression of VEGF and has been first choice of treating infantile hemangioma, the most common tumor of infancy. There are some pilot studies suggesting that the administration of oral propranolol is effective in counteracting the progression of ROP in patients without operation indication. Nevertheless that safety is a concern, for oral propranolol may result in associated complications and side effects such as bradycardia, hypotension, injury of cerebrum growth and olfactory.

Recently a research of eye drop propranolol in a mouse model of oxygen-induced retinopathy (OIR) has shown that propranolol was still effective in inhibiting angiogenic processes, indicating that local administration is equally effective.

The purpose of this study is to evaluate safety and efficacy of oral/local propranolol in preterm newborns with early phase of retinopathy of prematurity (ROP).The study will be followed up for a period of time, observing the development of optic and nerve system complications to further confirm the efficacy of propranolol to ROP treatment, which can provide theoretical basis for the futher clinical application of the drug in ROP.

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborns (birth weight less than 1500g) with stage 1/2 ROP in Zone 2 or 3 without plus
* A signed parental informed consent

Exclusion Criteria:

* Newborns with heart failure
* Newborns with recurrent bradycardia (heart rate < 90 beat per minute)
* Newborns with second or third degree atrioventricular block
* Newborns with congenital cardiovascular anomalies, except for persistent ductus arteriosus, patent foramen ovale and small ventricular septal defects
* Newborns with hypotension
* Newborns with renal failure
* Newborns with actual cerebral haemorrhage
* Newborns with other diseases which contraindicate the use of beta-adrenoreceptor blockers.
* Newborns with a more severe stage of ROP than stage 2 or in Zone 1

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-03 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of newborns who have ROP progression | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who need surgical treatment | participants will be followed for the duration of hospital stay, an expected average of 2 months
Number of newborns who have side effects | participants will be followed for the duration of hospital stay, an expected average of 2 months
Plasma concentrations of propranolol at the steady state measured by dried blood spots | 10th day of treatment

SECONDARY OUTCOMES:
visual assessment of enrolled newborns | about 12 months
Scores of Gesell development scale of enrolled newborns | about 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Nie, Doctor, Principal Investigator — Guangdong Women and Children Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zin A, Gole GA. Retinopathy of prematurity-incidence today. Clin Perinatol. 2013 Jun;40(2):185-200. doi: 10.1016/j.clp.2013.02.001. PMID 23719304
- [Background] Fierson WM; American Academy of Pediatrics Section on Ophthalmology; American Academy of Ophthalmology; American Association for Pediatric Ophthalmology and Strabismus; American Association of Certified Orthoptists. Screening examination of premature infants for retinopathy of prematurity. Pediatrics. 2013 Jan;131(1):189-95. doi: 10.1542/peds.2012-2996. Epub 2012 Dec 31. PMID 23277315
- [Background] Filippi L, Cavallaro G, Bagnoli P, Dal Monte M, Fiorini P, Donzelli G, Tinelli F, Araimo G, Cristofori G, la Marca G, Della Bona ML, La Torre A, Fortunato P, Furlanetto S, Osnaghi S, Mosca F. Oral propranolol for retinopathy of prematurity: risks, safety concerns, and perspectives. J Pediatr. 2013 Dec;163(6):1570-1577.e6. doi: 10.1016/j.jpeds.2013.07.049. Epub 2013 Sep 18. PMID 24054431
- [Background] Dal Monte M, Casini G, la Marca G, Isacchi B, Filippi L, Bagnoli P. Eye drop propranolol administration promotes the recovery of oxygen-induced retinopathy in mice. Exp Eye Res. 2013 Jun;111:27-35. doi: 10.1016/j.exer.2013.03.013. Epub 2013 Mar 23. PMID 23528535
- See also: Drug Information — https://druginfo.nlm.nih.gov/drugportal/name/propranolol